CLINICAL TRIAL: NCT04780087
Title: Experiences by Pregnant Power Athletes, and Health Related Outcomes in Mother and Infants, After Resistance Exercise Training During Pregnancy
Brief Title: Pregnant Women Doing Resistance Exercise Training
Acronym: PREG_RET
Status: Completed | Type: Observational
Sponsor: Ostfold University College (Other)
Responsible Party: Principal Investigator, Therese Fostervold Mathisen, Associate Professor, Ostfold University College
Other Study IDs: 170066
Record Dates: First submitted 2020-10-10; First posted 2021-03-03 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; Powerlifting; Weightlifting; Female athlete; Fertility; Delivery; Maternity leave; Resistance exercise training

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Weight lifting women: Experienced resistance exercise trained and pregnant women
- Reference women: Physically active pregnant women (not experienced with free weight lifting)

SUMMARY:
Despite the increase in numbers of women who engage in heavy, free-weight resistance exercise training (e.g. powerlifting, weightlifting, cross fit), the knowledge on how such exercise may affect fertility, pregnancy and birth outcomes is poor. Based on observational and associational studies of pregnant women in labour, recommendations are not to lift more than 11 kg in external load after mid-term, or to lift more than a total of 100 kg during a day. Ignoring such recommendations is associated to increased risk of miscarriage and preeclampsia, and of low birthweight and premature birth, respectively. As such, fit women who continue to exercise during pregnancy, are met with scepticism and warnings, resulting in shame and insecurity. Such attitudes may also result in physical inactivity during pregnancy, being on the contrary of what is recommended for a healthy pregnancy and delivery. Elite athletes may additionally be deprived from an early return to sport if not being able to keep exercise intensity close to pre-pregnancy period. With poor knowledge on how fit, strong women respond to high external loads during pregnancy exercise, recommendations are to follow the general guidelines.

The aim of this observational study, is to explore how regular resistance exercise training may affect fertility, and how high external loads in resistance exercise training during pregnancy in resistance trained women affect; a)their pregnancy and birth outcome, and b)health of the women and their children up to 12 months post-delivery.

DETAILED DESCRIPTION:
Pregnant women who are experienced in heavy, free-weight resistance exercise training, and who choose to continue their exercise regimes during pregnancy, are recruited in social media to regularly respond to an online questionnaire on personal health, foetus development, and the newborn child health.

A reference group of pregnant women being regularly physical active (still not lifting free weights of high loads) are concurrently recruited.

All will respond to questionnaire at mid-term, and week 23, 30 and 40 of pregnancy. During maternity leave the women will be asked to respond to questionnaires at 1 month, 3 months, 6 months and 12 months post-delivery.

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant
* Group of interest: Being experienced with heavy, free-weight resistance exercise training, and aiming to continue exercise at comparable level during pregnancy
* Reference group: being regularly physical active before pregnancy (i.e. at least 2 work- outs per week), but not experienced in heavy, free-weight resistance exercise training

Exclusion Criteria:

* Any known metabolic condition or contraindication on doing physical activity during pregnancy (i.e. miscarriages, bleedings).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Based on sex, as this study evaluates the effects from resistance exercise training on pregnancy outcomes
Study Population: Women included in "group of interest" are pregnant women who are experienced in heavy, free-weigth resistance exercise training (i.e. powerlifter, weightlifter, cross fit) who aim to continue exercise training during pregnancy.
  Reference group are pregnant women with no experience in heavy, free-weight resistance exercise, but who are regurlarly physically active in any sport activity (at least 2 times per week), and who aim to continue to exercise during pregnancy.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Delivery week | At delivery time
  The selfreported pregnancy week for delivery
Delivery method | At delivery time
  Participants report the method for delivery, choosing from natural delivery, delivery with assistance (e.g. birth forceps, vacuum delivery), caesarean section.
Pregnancy complications at week 23 | During pregnancy up to week 23
  Number of participants who report any complications during pregnancy, choosing from a list of alternatives (yes/no) (preeclampsia, nausea, fatigue, low back pain, pelvic pain, constipation, mood swings, birth anxiety, gestational depression, anemia, hypertension, pregnancy diabetes, foetus growth retardation)
Pregnancy complications at week 30 | Pregnancy week 23 to 30
  Number of participants who report any complications during pregnancy, choosing from a list of alternatives (yes/no) (preeclampsia, nausea, fatigue, low back pain, pelvic pain, constipation, mood swings, birth anxiety, gestational depression, anemia, hypertension, pregnancy diabetes, foetus growth retardation)
Pregnancy complications at week 40 | Pregnancy week 30 to 40
  Number of participants who report any complications during pregnancy, choosing from a list of alternatives (yes/no) (preeclampsia, nausea, fatigue, low back pain, pelvic pain, constipation, mood swings, birth anxiety, gestational depression, anemia, hypertension, pregnancy diabetes, foetus growth retardation)
Childs weight at birth | At delivery time
  The weight of the child
Childs length at birth | At delivery time
  The length of the child
Apgar score 5 minutes | At delivery time (5 minutes post-delivery)
  The Apgar score 5 minutes post-delivery. This test checks a baby's heart rate, muscle tone, and other signs to see if extra medical care or emergency care is needed. The test is usually given twice: once at 1 minute after birth, and again at 5 minutes after birth. Scores below 4 indicates need for lifesaving measures, and higher scores indicates better health.
Miscarriage | Previous and up to October 2023
  Number of miscarriages
Urinary incontinence before pregnancy | Any experience before pregnancy
  Number of participants reporting any challenges with urinary incontinence, and if it occurs; if it is only during increased abdominal pressure (coughing, laughing), or heavy lifting (choosing from a list of "always", only during increased abdominal pressure, only during lifting of heavy load)
Urinary incontinence during pregnancy | At pregnancy week 23, 30 and 40
  Number of participants reporting any urinary incontinence, and if it occurs; if it is only during increased abdominal pressure (coughing, laughing), or heavy lifting (choosing from a list of "always", only during increased abdominal pressure, only during lifting of heavy load)
Urinary incontinence after delivery | Post-delivery: 1 month-, 3months-, 6 months- and 12 months
  Number of participants reporting any urinary incontinence, and if it occurs; if it is only during increased abdominal pressure (coughing, laughing), or heavy lifting (choosing from a list of "always", only during increased abdominal pressure, only during lifting of heavy load)
Anal insufficiency before pregnancy | Any experience before pregnancy
  Number of participants reporting any challenges with fecal incontinence
Anal insufficiency during pregnancy | At pregnancy week 23, 30 and 40
  Number of participants reporting any challenges with fecal incontinence
Anal insufficiency after delivery | Post-delivery: 1 month-, 3months-, 6 months- and 12 months
  Number of participants reporting any fecal incontinence and if it has worsened after giving birth
Injuries during pregnancy up to week 23 | During pregnancy up to week 23
  Number of participants reporting on any exercise related injuries occuring during pregnancy, choosing from a list of anatomical locations
Injuries during pregnancy, up to week 30 | Pregnancy week 23 to 30
  Number of participants reporting on any exercise related injuries occuring during pregnancy, choosing from a list of anatomical locations
Injuries during pregnancy, up to week 40 | Pregnancy week 30 to 40
  Number of participants reporting on any exercise related injuries occuring during pregnancy, choosing from a list of anatomical locations (yes/no)
Analgesic during delivery | At delivery time
  Number of participants reporting use of analgesic during delivery, and what type of analgesic (e.g. nitrous oxide, epidural)

SECONDARY OUTCOMES:
Body weight at week 23 | Pregnancy week 23
  Participants report on body weight changes during pregnancy
Body weight at week 30 | Pregnancy week 30
  Participants report on body weight changes during pregnancy
Body weight at week 40 | Pregnancy week 40
  Participants report on body weight changes during pregnancy
Body weight post-delivery, 1month | Postpartum, 1 month after delivery
  Participants report on body weight changes after pregnancy
Body weight post-delivery, 3 months | Postpartum, 3 months after delivery
  Participants report on body weight changes after pregnancy
Body weight post-delivery, 6 months | Postpartum, 6 months after delivery
  Participants report on body weight changes after pregnancy
Body weight post-delivery, 12 months | Postpartum, 12 months after delivery
  Participants report on body weight changes after pregnancy
Changes in external loads used in exercise training | During pregnancy
  Participants report on changes in external loads used in exercise during pregnancy (% of normal loading used pre-pregnancy)
Changes in external loads used in exercise training, up to week 23 | During pregnancy, week 23
  Participants report on changes in external loads used in exercise during pregnancy (% of normal loading used pre-pregnancy)
Changes in external loads used in exercise training | Post-delivery: 1 month-, 3months-, 6 months- and 12 months
  Participants report on changes in external loads used in exercise after pregnancy (% of normal loading used pre-pregnancy)
Changes in exercise volume during pregnancy, up to week 23 | During pregnancy, week 23
  Participants report on changes in exercise volume (number of sessions per week) during pregnancy
Changes in exercise volume during pregnancy, up to week 30 | During pregnancy, week 30
  Participants report on changes in exercise volume (number of sessions per week) during pregnancy
Changes in exercise volume during pregnancy, up to week 40 | During pregnancy, week 40
  Participants report on changes in exercise volume (number of sessions per week) during pregnancy
Changes in exercise volume after pregnancy | Post-delivery: 1 month-, 3months-, 6 months- and 12 months
  Participants report on changes in exercise volume (number of sessions per week) after pregnancy
Injuries from exercise during maternity leave | Post-delivery: 1 month-, 3months-, 6 months- and 12 months
  Reporting on any exercise related injuries occuring during maternity leave (up to 12 months post-delivery), choosing from a list of anatomical locations
Fertility | Before pregnancy
  Reports on any fertility problems or use of fertility techniques in order to become pregnant
Bloodpressure | At pregnancy week 23, 30 and 40, and at 1 month-, 3months-, 6 months- and 12 months postdelivery,
  Bloodpressure measures, and numbers above/below clinical cut offs (having hypo-or hypertension)
Symphysis-fundus measure | At pregnancy week 23, 30 and 40
  symphysis fundus measure during pregnancy; as a measure for growth of the fetus, evaluated according to national/international standards

OTHER OUTCOMES:
Use of supplements | At pregnancy week 23, 30 and 40, and at 1 month-, 3months-, 6 months- and 12 months postdelivery,
  Number of participants reporting use of dietary supplements, and what kind of supplements
Use of caffein (coffee, energydrinks, sodawater) | At pregnancy week 23, 30 and 40, and at 1 month-, 3months-, 6 months- and 12 months postdelivery,
  Number of participants reporting use of caffein, and in what doses per day
Intake of alcohol | At pregnancy week 23, 30 and 40, and at 1 month-, 3months-, 6 months- and 12 months postdelivery,
  Number of participants reporting intake of alcohol, and how regularly (choosing between no, daily, weekly, monthly)
Use of tobacco/cigarettes or snus | At pregnancy week 23, 30 and 40, and at 1 month-, 3months-, 6 months- and 12 months postdelivery,
  Number of participants reporting any use
Use of any prescribed drugs | At pregnancy week 23, 30 and 40, and at 1 month-, 3months-, 6 months- and 12 months postdelivery,
  Number of participants reporting any use, and what type of drug

CONTACTS AND LOCATIONS:
Overall Officials: Therese F Mathisen, PhD, Principal Investigator — Østfold University College
Locations (1):
- Therese Fostervold Mathisen, Fredrikstad, Norway

IPD SHARING:
Plan to Share IPD: No
Data are kept within the research group